CLINICAL TRIAL: NCT07055074
Title: Evaluation of Hemodynamic Changes Using Different Intra-Abdominal Pressures for Laparoscopic Cholecystectomy Under General Anesthesia
Brief Title: Evaluation of Hemodynamic Changes Using Different IAP for LC Under General Anesthesia
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHSW/Batch-Fall23/918
Record Dates: First submitted 2025-06-26; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Laparocele

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low Pressure Pneumoperitoneum
  Interventions: Diagnostic Test: Low Pressure Pneumoperitoneum
- Medium Pressure Pneumoperitoneum
  Interventions: Diagnostic Test: Medium Pressure Pneumoperitoneum

INTERVENTIONS:
Diagnostic Test: Low Pressure Pneumoperitoneum — Low Pressure Pneumoperitoneum (8-10 mmHg) Details: CO₂ insufflation to 8-10 mmHg IAP, continuous monitoring, measurement at baseline, insufflation, and desufflation.
  Groups: Low Pressure Pneumoperitoneum
Diagnostic Test: Medium Pressure Pneumoperitoneum — Medium Pressure Pneumoperitoneum (12-14 mmHg) Details: CO₂ insufflation to 12-14 mmHg IAP, parameters measured at key intervals, standard general anesthesia used. High Pressure Pneumoperitoneum (15-20 mmHg) Details: Standard high-pressure technique, monitoring of hemodynamic and respiratory parameters.
  Groups: Medium Pressure Pneumoperitoneum

SUMMARY:
This cross-sectional observational study aims to evaluate the hemodynamic changes induced by different intra-abdominal pressures (IAP) during laparoscopic cholecystectomy under general anesthesia.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy, a minimally invasive surgery, requires CO₂ insufflation to create a pneumoperitoneum, which alters intra-abdominal pressure and can affect cardiovascular and respiratory stability. This study assesses how varying IAP levels (8-10 mmHg, 12-14 mmHg, and 15-20 mmHg) influence heart rate, blood pressure, oxygen saturation, respiratory rate, and end-tidal CO₂.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic cholecystectomy under general anesthesia
* Age between 18-60 years
* ASA physical status I-II
* Provided informed consent

Exclusion Criteria:

* History of cardiovascular or respiratory diseases or other Significant comorbidities affecting hemodynamic stability.
* Pregnant patients
* Allergies to anesthetic agents

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Hemodynamic stability, intra-abdominal pressure effects, physiological stress during laparoscopic cholecystectomy, cardiovascular and respiratory responses under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Self Administered Questioner | 12 Months
  Self-Administered Questionnaire for taking different values

CONTACTS AND LOCATIONS:
Locations (1):
- Pakistan Surgical Center, G9/4, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No